CLINICAL TRIAL: NCT02791048
Title: Evaluation of the Effectiveness of Music Therapy in Improving the Quality of Life of Palliative Care Patients: a Randomised Controlled Pilot and Feasibility Study
Brief Title: Music Therapy for Palliative Care Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University, Belfast (Other)
Collaborators: Marie Curie Hospice, Belfast (Other); Every Day Harmony Music Therapy (Northern Ireland Music Therapy Trust) (Unknown)
Responsible Party: Principal Investigator, Dr Joanne Reid, Dr, Queen's University, Belfast
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B16/27
Record Dates: First submitted 2016-05-25; First posted 2016-06-06 (Estimated); Last update posted 2019-03-21 (Actual); Status verified 2019-03

CONDITIONS: Palliative Care
MeSH Terms: interventions — Music Therapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental Group (Experimental): Music therapy for up to 45 minutes twice a week for three weeks, in addition to usual care from the hospice multidisciplinary team.
  Interventions: Behavioral: Music therapy
- Control Group (No Intervention): Usual care only from the hospice multidisciplinary team. The dose and frequency of usual care will be as deemed appropriate by the hospice practitioner in charge of their treatment.

INTERVENTIONS:
Behavioral: Music therapy — Music therapy is a clinical intervention conducted by qualified therapists who use shared music-making and improvisation to engage and interact with the client (s) in order to work towards specific therapeutic objectives.
  This is the aim of sessions, rather than the teaching or utilising of any musical skills, and clients do not have to have any prior musical training or experience whatsoever in order to participate in and benefit from music therapy. The intervention is client-led and the therapist will guide the patient in a range of strategies and activities appropriate to the therapeutic aims in place. Sessions can be individual, or family members can also be involved if appropriate and desired.
  Arms: Experimental Group

SUMMARY:
This study aims to find out if music therapy is effective in improving the quality of life of palliative care patients. It will do this by comparing palliative care patients who receive music therapy with those who do not receive music therapy.

DETAILED DESCRIPTION:
Quality of life (QOL) is very important for palliative care patients, and includes the physical, psychological, social, and spiritual aspects of a patient's life. Music therapy is often used to help palliative care patients and there is some evidence that music therapy helps improve their quality of life, especially in relation to reducing levels of pain. Many palliative care patients and their families have also said that music therapy is helpful. However, more research is needed to help healthcare providers and funders decide if music therapy really is a useful treatment for patients receiving palliative care.

ELIGIBILITY:
Inclusion Criteria:

Only patients deemed able to engage with interactive music therapy will be invited to join the study. Eligibility will be assessed by a clinician during inpatient admission using the Eastern Cooperative Oncology Group (ECOG) scale and the Abbreviated Mental Test (AMT).

* Patients will be eligible if they have an ECOG performance status of 0, 1, 2 or 3 (0 indicating the patient is asymptomatic, 1 the patient is symptomatic but fully ambulatory, 2 the patient is symptomatic and confined to bed for less than 50% of the day, and 3 the patient is symptomatic and confined to bed for more than 50% of the day)) indicating they are able to engage with interactive music therapy. - Eligible patients will also have a score of 7 or more on the AMT, indicating they are capable of providing meaningful informed consent and accurate responses to the study's primary outcome measurement tool.
* Patients with communication difficulties will also be eligible if they are able to indicate their responses to the questionnaire.
* Musical skills are not required. Prior musical skills will not lead to exclusion from the study. The patient must freely consent to participation following receipt of information about the trial.

Exclusion Criteria:

* Patients will be excluded from the study if they have an ECOG performance status of 4 (4 indicating the patient is severely symptomatic and completely bedridden) or a score of 6 or less on the AMT, indicating they may not be capable of providing fully informed consent or accurate responses to the study's primary outcome measurement tool.
* Participants who decide not to consent will be excluded from the trial. Patients will be assured that this decision will have no implications for the care that they receive.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2016-04; Primary Completion 2017-06 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Quality of life | Up to 12 months
  Quality of life will be measured using the McGill Quality of Life Questionnaire: MQOL (Cohen et al., 1995), which contains 17 items, and has been shown to have the best clinimetric quality rating, content validity, construct validity and internal consistency of reviewed quality of life questionnaires in a systematic review (Albers et al., 2010). Out of 29 instruments evaluated, only the MQOL demonstrated good reliability. However, the McGill Quality of Life Questionnaire-Cardiff Short Form (MQOL-CSF: 8 items) (Pratheepawanit et al., 1999), will be considered as an alternative for the main trial if the former instrument is found to place undue burden on respondents. An analysis of the feasibility, reliability and validity of the MQOL-CSF concluded 'that the MQOL-CSF is a feasible tool with favourable psychometric properties for routine HRQoL assessment in the palliative care population' (Lua et al., 2005: 1669).

SECONDARY OUTCOMES:
The effect of music therapy upon quality of life two weeks after completion of the music therapy course | Up to 12 months
  Quality of life will be measured using the McGill Quality of Life Questionnaire: MQOL (Cohen et al., 1995), which contains 17 items, and has been shown to have the best clinimetric quality rating, content validity, construct validity and internal consistency of reviewed quality of life questionnaires in a systematic review (Albers et al., 2010). Out of 29 instruments evaluated, only the MQOL demonstrated good reliability. However, the McGill Quality of Life Questionnaire-Cardiff Short Form (MQOL-CSF: 8 items) (Pratheepawanit et al., 1999), will be considered as an alternative for the main trial if the former instrument is found to place undue burden on respondents. An analysis of the feasibility, reliability and validity of the MQOL-CSF concluded 'that the MQOL-CSF is a feasible tool with favourable psychometric properties for routine HRQoL assessment in the palliative care population' (Lua et al., 2005: 1669).
The effect of music therapy upon inter-familial communication | Up to 12 months
  In the absence of a validated tool to measure this outcome the investigators propose to use qualitative interviewing of family/carers to ascertain if music therapy altered the quality of communication between them and patients.
The effect of contextual factors upon the implementation and sustainability of music therapy in a palliative care setting | Up to 12 months
  Marie Curie Hospice employees with a direct patient care role will be invited to take part in a focus group. The aim is to develop an integrated outcome and process evaluation framework to advance theoretical understanding of what components of music therapy work best, for whom, and in what circumstances.

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Reid, Dr, Principal Investigator — School of Nursing and Midwifery, Queen's University Belfast
Locations (1):
- Marie Curie Hospice, Belfast, Co. Antrim, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Porter S, McConnell T, Graham-Wisener L, Regan J, McKeown M, Kirkwood J, Clarke M, Gardner E, Dorman S, McGrillen K, Reid J. A randomised controlled pilot and feasibility study of music therapy for improving the quality of life of hospice inpatients. BMC Palliat Care. 2018 Nov 27;17(1):125. doi: 10.1186/s12904-018-0378-1. PMID 30482192
- [Derived] McConnell T, Graham-Wisener L, Regan J, McKeown M, Kirkwood J, Hughes N, Clarke M, Leitch J, McGrillen K, Porter S. Evaluation of the effectiveness of music therapy in improving the quality of life of palliative care patients: a randomised controlled pilot and feasibility study. Pilot Feasibility Stud. 2016 Nov 29;2:70. doi: 10.1186/s40814-016-0111-x. eCollection 2016. PMID 27965885